CLINICAL TRIAL: NCT03921242
Title: Comparative Effectiveness of Metformin for Type 2 Diabetes With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 1809019555
Record Dates: First submitted 2019-04-08; First posted 2019-04-19 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — Metformin; Sulfonylurea Compounds; Dipeptidyl-Peptidase IV Inhibitors; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Metformin Cohort: Group of study participants having both Type 2 Diabetes and Chronic Kidney disease and meeting the study's inclusion criteria for whom metformin was prescribed at baseline for this first time in each patient's medical history.
  Interventions: Drug: Metformin
- Sulfonylurea Cohort: Group of study participants having both Type 2 Diabetes and Chronic Kidney disease and meeting the study's inclusion criteria for whom sulfonylurea was prescribed at baseline for this first time in each patient's medical history.
  Interventions: Drug: Sulfonylurea
- DPP4 Inhibitor Cohort: Group of study participants having both Type 2 Diabetes and Chronic Kidney disease and meeting the study's inclusion criteria for whom a DPP4 Inhibitor was prescribed at baseline for this first time in each patient's medical history.
  Interventions: Drug: DPP-4 inhibitor
- SGLT2 Inhibitor Cohort: Group of study participants having both Type 2 Diabetes and Chronic Kidney disease and meeting the study's inclusion criteria for whom an SGLT2 Inhibitor was prescribed at baseline for this first time in each patient's medical history.
  Interventions: Drug: SGLT2 inhibitor
- GLP1 Receptor Agonist Cohort: Group of study participants having both Type 2 Diabetes and Chronic Kidney disease and meeting the study's inclusion criteria for whom a GLP1 receptor agonist was prescribed at baseline for this first time in each patient's medical history.
  Interventions: Drug: GLP1 receptor agonist

INTERVENTIONS:
Drug: Metformin — Newly Initiated and regular metformin dosage as prescribed by each patient's medical care provider
  Groups: Metformin Cohort
Drug: Sulfonylurea — Newly initiated and regular sulfonylurea dosage as prescribed by each patient's medical care provider
  Groups: Sulfonylurea Cohort
Drug: DPP-4 inhibitor — Newly initiated and regular DPP-4 inhibitor dosage as prescribed by each patient's medical care provider
  Groups: DPP4 Inhibitor Cohort
Drug: SGLT2 inhibitor — Newly initiated and regular SGLT2 inhibitor dosage as prescribed by each patient's medical care provider
  Groups: SGLT2 Inhibitor Cohort
Drug: GLP1 receptor agonist — Newly initiated and regular GLP1 receptor agonist dosage as prescribed by each patient's medical care provider
  Groups: GLP1 Receptor Agonist Cohort

SUMMARY:
This is a proposal for a retrospective observational study of the safety of metformin use in patients with chronic kidney disease, compared to other commonly used diabetes drugs. It will be conducted using retrospective data from the New York City CDRN, Medicare administrate files, and New York State Medicaid administrative files, which will be linked and then deidentified prior to analysis.

DETAILED DESCRIPTION:
Specific aims are as follows:

Aim 1. For patients with Type 2 Diabetes Mellitus(T2DM) and Chronic Kidney Disease (CKD), compare metformin to alternative non-insulin diabetes drugs (sulfonylureas, DPP-4 inhibitors, GLP-1 receptor agonists, and SGLT-2 inhibitors)) with respect to the key safety outcome of severe hypoglycemia. The primary hypothesis is that metformin will be superior to sulfonylurea in terms of severe hypoglycemia rates, and non-inferior to DPP-4 inhibitors. Secondary outcomes will include hospitalization for acidosis, hospitalization for hyperglycemia, acute myocardial infarction, stroke, heart failure hospitalization, and heart failure emergency room visit.

Aim 2. For patients with T2DM and CKD, compare metformin to alternative non-insulin diabetes drugs with respect to HbA1c reduction. The primary hypothesis is that metformin will be superior to DPP-4 inhibitors and non-inferior to sulfonylureas for HbA1c reduction (i.e., improvement in blood sugar). Secondary outcomes will include change in body-mass index (BMI) and kidney function, non-persistence to treatment, and progression to insulin use.

Aim 3. Examine the heterogeneity of treatment effects on hypoglycemia risk and HbA1c response across patient subgroups. The primary hypothesis is that metformin's advantages will be more pronounced in more severe CKD.

Aim 4 (data completeness): Using the linked Medicare-CDRN dataset, assess completeness of CDRN data for drugs and hospitalization among Medicare recipients. Specifically, we will use Medicare data from 2013-2016 as a gold standard and assess the sensitivity, specificity, negative predictive value (NPV), and positive predictive value (PPV) of INSIGHT CDRN data from those years in identifying hospitalizations and prevalent diabetes drug use among Medicare patients with T2DM (type 2 diabetes mellitus), and develop and validate an algorithm to identify patients for whom NPV and PPV for hospitalizations and all major diabetes drug classes exceed 80%. We hypothesize that such an algorithm will identify a population of a quarter of eligible Medicare patients in the CDRN who meet or exceed these standards for completeness of data.

Aim 5. Conduct a cohort study to test the hypothesis that poorly controlled baseline HbA1c is not independently associated with the primary outcome (hospitalization with COVID). Primary analysis will be restricted to Medicare patients identified by aim 1 as likely to surpass 80% NPV and PPV for the primary outcome. A finding that HbA1c is not associated with worse outcomes would support relaxing glycemic targets during the pandemic when this allows patients to avoid unnecessary risks associated with aggressive treatment, monitoring, and exposure to the health care system.

Aim 6: Conduct a comparative cohort study to test the null hypothesis that metformin, SGLT-2 inhibitors, DPP-4 inhibitors, GLP-1 receptor agonists, and sulfonylureas do not have class-specific effects on the primary outcome. Primary analysis will be restricted to Medicare patients identified by aim 1 as likely to surpass 80% NPV and PPV both for the primary outcome and exposure to the drug of interest. Two sub-hypotheses would be of special interest: if SGLT-2 inhibitors are associated with increased risk, this would support suggestions that they be temporarily stopped in high risk patients; if DPP-4 inhibitors are associated with decreased risk, this would argue for prospective research into this class as protective agents.

ELIGIBILITY:
Inclusion Criteria:

* A coded inpatient or outpatient T2DM diagnosis (ICD9/ICD10) and an antidiabetic medication prescription within the 90 days following the diagnosis date (CP1); a coded T2DM diagnosis and an outpatient glycolated hemoglobin (HbA1C) value≥6.5% within 90 days before or after the diagnosis date (CP2); or any antidiabetic medication prescription within 90 days before or after an outpatient HbA1C value ≥6.5% (CP3).
* New use of a medication of interest (metformin, sulfonylurea, DPP4 inhibitor, SGLT2 inhibitor, or GLP1 receptor agonist
* Estimated glomerular filtration rate (eGFR) of less than 60 ml/min within the month prior to the new medication

Exclusion Criteria:

* Coded diagnoses of gestational diabetes
* Coded diagnoses of prediabetes
* Coded diagnoses of type 1 diabetes
* Evidence of a positive beta human chorionic gonadotropin test as a marker for pregnancy during the 90 days before or after the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: EHR data from two data sources (NYC and Mid-South CDRN's) will be linked to insurance claims data to identify adult patients (age > 18) with T2DM and CKD, who are initiating metformin or one of the comparator drugs. Also, participants will further be required to have at least one prescription for metformin, sulfonylurea, or DPP-4 inhibitor; at least 6 months preceding that prescription in which none of those drugs are used; and an eGFR within 1 month prior to the index date (the date on which the drug of interest is started) of < 60 mL/min
Sampling Method: Non-Probability Sample
Enrollment: 4888 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Severe Hypoglycemia Assessed from EMR | 18 Months
  Comparing the time-to event outcomes between metformin and other index exposures. Severe Hypoglycemic events are defined as events resulting in emergency room, observation, or inpatient visits where hypoglycemia is the primary diagnosis
Difference in Glycosylated Hemoglobin (HbA1c) level (mmol/mol) | 24 Months
  Comparing the change in HbA1c in the metformin-initiator cohort to the changes reported in the sulfonylurea- and DPP4-I-initiator cohorts at 3-9 months following baseline. HbA1c will be measured in mmol/mol.
Heterogeneity of Treatment Effect Via Pre-specified Sub-Group Analyses | 25 Months
  Determine the extent of heterogeneity in treatment effect through the stratification of the sample population by covariate subgroups (age, sex, BMI, race; baseline history of CVD, liver disease, and heart failure; specific sulfonylurea or DPP-4 inhibitor, and levels of renal function and metformin dose as time-varying covariates) and through the use of machine learning techniques.

SECONDARY OUTCOMES:
Incidence of acidosis, hospitalization for hyperglycemia, acute myocardial infarction, stroke, heart failure hospitalization, and heart failure emergency room visits | 18 Months
  Comparing the time-to event outcomes between the metformin and other index exposure cohorts in terms of occurrences of acidosis, hospitalizations for hyperglycemia, acute myocardial infarction, stroke, heart failure hospitalizations, and heart failure emergency room visits
Difference in Glycosylated Hemoglobin (HbA1c) level (mmol/mol) | 24 Months
  Comparing the change in HbA1c in the metformin-initiator cohort to the changes reported in the sulfonylurea- and DPP4-I-initiator cohorts at 12-24 months following baseline. HbA1c will be measured in mmol/mol.
Difference in Body-Mass Index Assessed From EMR (BMI) (kg/m2) | 24 Months
  Comparing the change in body-mass index (BMI) in the metformin-initiator cohort to the changes reported in the sulfonylurea- and DPP4-I-initiator cohorts. BMI will be measured in kg/m2.
Difference in Laboratory-Measured eGFR (mL/min) | 24 Months
  Comparing the change in eGFR in the metformin-initiator cohort to the changes reported in the sulfonylurea- and DPP4-I-initiator cohorts. eGFR will be measured in mL/min.

CONTACTS AND LOCATIONS:
Overall Officials: Alvin Mushlin, Principal Investigator — Weill Cornell Medical College/Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - University of North Carolina, Chapel Hill, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No